CLINICAL TRIAL: NCT03835117
Title: Effect of a Wide Spectrum Nutritional Supplement on Mitochondrial Function in Children With Autism Spectrum Disorder (ASD)
Brief Title: Effect of a Wide Spectrum Nutritional Supplement on Mitochondrial Function in Children With Autism Spectrum Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rossignol Medical Center (Other)
Collaborators: Southwest Autism Research & Resource Center (Other)
Responsible Party: Principal Investigator, Richard Frye, Director of Research, Rossignol Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MITO
Record Dates: First submitted 2019-02-05; First posted 2019-02-08 (Actual); Results first posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-04

CONDITIONS: Autism Spectrum Disorder
Keywords: Mitochondrial Dysfunction
MeSH Terms: conditions — Autism Spectrum Disorder; Mitochondrial Diseases

STUDY DESIGN:
Intervention Model Description: Prospective Randomized 12-week Double-Blind Placebo-Controlled Cross-over
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Wide-spectrum nutritional supplement (Experimental): The Wide-spectrum nutritional supplement used will be a combination of NeuroNeeds: SpectrumNeeds and QNeeds. Weight based dosing will be used. The daily serving size will be divided into two oral daily doses in the form of a powder which can be mixed into liquid or food. Together, there are 34 different dietary supplements in the products. Except for ubiquinol, all of these nutrients are provided in a powder form in SpectrumNeeds. Ubiquinol is provided separately in QNeeds gel capsules. These capsules can be swallowed whole, or cut with scissors and the contents squeezed out and added to SpectrumNeeds just before ingestion.
  Interventions: Drug: Wide-spectrum nutritional supplement
- Placebo control (Placebo Comparator): Participants randomized to receive placebo will take placebo in an oral form divided into powder and a gel capsule in the same manner as treatment. For the second phase of the cross over, participants will be part of the opposite group they were assigned to in Phase I (Placebo or Treatment). Quantities for placebo or treatment will match across phases for each subject, utilizing the same weight based dosing.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Wide-spectrum nutritional supplement — Comprehensive powder with 33 dietary supplements and 1 dietary supplement via gel capsule.
  Other Names: NeuroNeeds: Spectrum Needs, NeuroNeeds:Q Needs
  Arms: Wide-spectrum nutritional supplement
Other: Placebo — Inactive placebo comparator
  Arms: Placebo control

SUMMARY:
The objective of this study is to evaluate the metabolic effects of a comprehensive wide-spectrum supplement for children with ASD to determine whether it physiologically targets mitochondrial pathways known to be abnormal in children with ASD.The intervention is a commonly used wide-spectrum nutritional supplement, which is theoretically designed to normalize mitochondrial function. The investigators aim to determine if the supplement does have the hypothesized effect on physiology in individuals with ASD. The investigator will enroll up to 50 children, aged 4 to 14 years of age with confirmed ASD and mitochondrial dysfunction, and participation will last 26 weeks.

DETAILED DESCRIPTION:
Autism spectrum disorder (ASD) is a heterogeneous neurodevelopmental disorder often with life-long consequences that affects young children during critical developmental periods. The Centers for Disease Control estimates that ASD affects as many as 17 per 1000 children (1 in 59) in the United States suggesting that the prevalence is higher than previous estimates.Despite the dramatic rise in the detected prevalence of ASD over the past two decades, there is no effective medical treatment for core ASD symptoms (social communication and repetitive behavior), the closely associated problem of language impairment, or the underlying pathophysiology of ASD. Currently, the only accepted treatment for core ASD symptoms is behavior therapy, which may entail intensive one-on-one treatment over several years.

The primary aims of this study are to evaluate the effect of a wide-spectrum nutritional supplement on mitochondrial function in individuals with ASD. Participants entered into the trial will have abnormalities in mitochondrial function that are known to be associated with ASD (approximately 50+% of children with ASD) but are not diagnostic of mitochondrial disease. The investigators hypothesize that nutritional supplements designed for children with ASD have a physiological action of normalizing mitochondrial function and cellular physiology throughout the body.

To test whether the targeted nutritional supplement is superior to placebo, the investigators will study 50 children, between the ages of 4 years to 14 years, with confirmed ASD and known abnormal variations in mitochondrial at baseline. Participants will be randomly assigned to receive active treatment or placebo for 12-weeks under double-blind conditions and at the end of the 12 weeks switch to the opposite condition after a 2-week wash out period. Mitochondrial function will be measured at baseline and after each treatment arm in order to determine if the supplement positively influences cellular biochemistry. The investigator will also evaluate the effectiveness of the supplement on core and associated ASD symptoms using several behaviors assessments.

ELIGIBILITY:
Inclusion Criteria:

* Weight ≥ 15 kg and ≤ 100kg;
* DSM-5 diagnosis of Autism Spectrum Disorder as established by formal clinical assessment which includes a gold-standard tool such as the Autism Diagnostic Observational Schedule.
* Current Clinical Global Impression Severity score ≥ 4
* Stable educational and therapy plan (one month) with no planned changes in the intensity of treatment for 12 weeks.
* English is spoken in the home and at least one parent is able to read, write and speak English.
* Stable medication (no changes in past 6 weeks and no planned changes for the study duration.
* Electron Transport Chain Complex (I, II, III, IV) or Citrate Synthase Activity which is >= 2.0 Standard Deviation Above or Below Average (outside the normal range)

Exclusion Criteria:

* Presence of serious behavioral problems (tantrums, aggression, self-injury) for which another treatment is warranted.
* Current Clinical Global Impression Severity score < 7 (Extremely Ill)
* Significant medical condition by history or by physical examination or lab tests that would be incompatible with the treatment.
* Children taking anticonvulsant medication for seizures or active epilepsy.
* Diagnosis of Mitochondrial Disease

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard E Frye, MD, PhD, Principal Investigator — Rossignol Medical Center, Phoenix AZ
Locations (1):
- Southwestern Research & Resource Center, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Delhey LM, Nur Kilinc E, Yin L, Slattery JC, Tippett ML, Rose S, Bennuri SC, Kahler SG, Damle S, Legido A, Goldenthal MJ, Frye RE. The Effect of Mitochondrial Supplements on Mitochondrial Activity in Children with Autism Spectrum Disorder. J Clin Med. 2017 Feb 13;6(2):18. doi: 10.3390/jcm6020018. PMID 28208802
- [Background] Rose S, Niyazov DM, Rossignol DA, Goldenthal M, Kahler SG, Frye RE. Clinical and Molecular Characteristics of Mitochondrial Dysfunction in Autism Spectrum Disorder. Mol Diagn Ther. 2018 Oct;22(5):571-593. doi: 10.1007/s40291-018-0352-x. PMID 30039193
- [Background] Frye RE, Rossignol DA. Treatments for biomedical abnormalities associated with autism spectrum disorder. Front Pediatr. 2014 Jun 27;2:66. doi: 10.3389/fped.2014.00066. eCollection 2014. PMID 25019065

RESULTS

PARTICIPANT FLOW:
Groups:
- Wide-spectrum Nutritional Supplement First: The Wide-spectrum nutritional supplement used will be a combination of NeuroNeeds: SpectrumNeeds and QNeeds. Weight based dosing will be used. The daily serving size will be divided into two oral daily doses in the form of a powder which can be mixed into liquid or food. Together, there are 34 different dietary supplements in the products. Except for ubiquinol, all of these nutrients are provided in a powder form in SpectrumNeeds. Ubiquinol is provided separately in QNeeds gel capsules. These capsules can be swallowed whole, or cut with scissors and the contents squeezed out and added to SpectrumNeeds just before ingestion.
  Wide-spectrum nutritional supplement: Comprehensive powder with 33 dietary supplements and 1 dietary supplement via gel capsule.
- Placebo Control First: Participants randomized to receive placebo will take placebo in an oral form divided into powder and a gel capsule in the same manner as treatment. For the second phase of the cross over, participants will be part of the opposite group they were assigned to in Phase I (Placebo or Treatment). Quantities for placebo or treatment will match across phases for each subject, utilizing the same weight based dosing.
  Placebo: Inactive placebo comparator
Period: Phase I - Week 1 to Week 12
Arm/Group | Wide-spectrum Nutritional Supplement First | Placebo Control First
Started | 7 | 9
Completed | 7 | 9
Not Completed | 0 | 0
Period: Phase II - Week 13- Week 24
Arm/Group | Wide-spectrum Nutritional Supplement First | Placebo Control First
Started | 7 | 9
Completed | 5 | 6
Not Completed | 2 | 3
Not completed — Lost to Follow-up | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Wide-spectrum Nutritional Supplement First | Placebo Control First | Total
Number analyzed (Participants) | 7 | 9 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.7 (4.1) | 9.0 (3.9) | 9.3 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 7 | 7 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 4 | 6 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 5 | 7 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 9 | 16

OUTCOME MEASURES:

1. Primary Outcome: Change in Mitochondrial Activity in Study Patients: Citrate Synthase
Description: Mitochondrial activity and redox metabolism at baseline and after the placebo and supplement arms of the study, as determined through laboratory assessment. Normal Range 4.4 to 22 with Mean and SD of 12.1 and 5.1. It is better to be within the normal range than outside of the normal range regardless of whether the value is higher or lower.
Time Frame: Before (Baseline), After Part I (Week 12), After Part 2 (Week 24)
Population: Results are for Placebo and Treatment arm. Flow is for which treatment given first.
Measure: Mean (Standard Deviation); unit: nmoles/min/mg protein
Arm/Group | Wide-spectrum Nutritional Supplement | Placebo Control
Number analyzed (Participants) | 16 | 16
nmoles/min/mg protein
  Before | 40.56 (16.64) | 29.09 (11.48)
  After | 27.41 (6.43) | 37.78 (16.89)

2. Primary Outcome: Change in Mitochondrial Activity in Study Patients: Complex I
Description: Mitochondrial activity and redox metabolism at baseline and after the placebo and supplement arms of the study, as determined through laboratory assessment. Normal range is 3.4 to 11.9 with a mean of 7.65. Outside of the normal range is worse regardless of whether it is above or below the normal range.
Time Frame: Before (Baseline), After Part I (Week 12), After Part 2 (Week 24)
Population: Results are for Placebo and Treatment arm. Flow is for which treatment given first.
Measure: Mean (Standard Deviation); unit: Ratio of Complex I to Citrate Synthase
Arm/Group | Wide-spectrum Nutritional Supplement | Placebo Control
Number analyzed (Participants) | 16 | 16
Ratio of Complex I to Citrate Synthase
  Before | 2.88 (1.37) | 3.31 (1.99)
  After | 2.98 (1.65) | 2.86 (0.93)

3. Primary Outcome: Change in Mitochondrial Activity in Study Patients: Complex II
Description: Mitochondrial activity and redox metabolism at baseline and after the placebo and supplement arms of the study, as determined through laboratory assessment. Normal Range (mean ±SD) 0.03 -- 0.35 (0.194 ±0.08). It is better to be within the normal range regardless of whether the value is above or below the normal range
Time Frame: Before (Baseline), After Part I (Week 12), After Part 2 (Week 24)
Population: Results are for Placebo and Treatment arm. Flow is for which treatment given first.
Measure: Mean (Standard Deviation); unit: Ratio of Complex II to Citrate Synthase
Arm/Group | Wide-spectrum Nutritional Supplement | Placebo Control
Number analyzed (Participants) | 16 | 16
Ratio of Complex II to Citrate Synthase
  Before | 0.10 (0.06) | 0.09 (0.05)
  After | 0.09 (0.06) | 0.09 (0.06)

4. Primary Outcome: Change in Mitochondrial Activity in Study Patients: Complex IV
Description: Mitochondrial activity and redox metabolism at baseline and after the placebo and supplement arms of the study, as determined through laboratory assessment. Normal Range (mean ±SD) 0.15 -- 0.6 (0.31 ±0.1). Better scores are inside the normal range regardless of if they are higher or lower.
Time Frame: Before (Baseline), After Part I (Week 12), After Part 2 (Week 24)
Population: Results are for Placebo and Treatment arm. Flow is for which treatment given first.
Measure: Mean (Standard Deviation); unit: Ratio of Complex IV to Citrate Synthase
Arm/Group | Wide-spectrum Nutritional Supplement | Placebo Control
Number analyzed (Participants) | 16 | 16
Ratio of Complex IV to Citrate Synthase
  Before | 0.18 (0.04) | 0.21 (0.07)
  After | 0.22 (0.04) | 0.17 (0.03)

5. Secondary Outcome: Change in the Childhood Autism Rating Scale (CARS) Score
Description: The Childhood Autism Rating Scale is a 15-item clinician-rated scale that measures the severity of core ASD symptoms of social communication and restricted and repetitive patterns of behavior, interests, or activities. Each item is scored on a 4 point scale of severity from 1 (None/Minimal) to 4 (Severe). Minimal score is 15 and maximal score is 60. The measure is the total score of the 15 items in which a score of 15-27.5 reflects minimal to no severity of symptoms, 28-33.5 reflects mild to moderate severity of symptoms, and a score of 34 or higher reflects severe symptoms. Lower scores are better.
Time Frame: Before (Baseline), After Part I (Week 12), After Part 2 (Week 24)
Measure: Mean (Standard Deviation); unit: CARS Scale Units
Arm/Group | Wide-spectrum Nutritional Supplement | Placebo Control
Number analyzed (Participants) | 16 | 16
CARS Scale Units
  Before | 34.2 (9.9) | 37.2 (6.8)
  After | 30.8 (10.7) | 32.2 (3.4)

6. Secondary Outcome: Change in the Clinical Global Impression Scale (CGI) Score
Description: The Clinical Global Impression - Severity scale (CGI-S) is a clinician rated 7-point measure of overall symptomatic severity of psychopathology. Scores range from 1 (Normal, not at all ill) through 4 (Moderately ill) to 7 (Among the most extremely ill patients). Lower scores are better.
Time Frame: Before (Baseline), After Part I (Week 12), After Part 2 (Week 24)
Measure: Mean (Standard Deviation); unit: Raw Score
Arm/Group | Wide-spectrum Nutritional Supplement | Placebo Control
Number analyzed (Participants) | 16 | 16
Raw Score
  Before | 4.5 (1.3) | 4.69 (1.1)
  After | 4.31 (1.4) | 4.31 (1.1)

7. Secondary Outcome: Change in the Children's Yale-Brown Obsessive Compulsive Scale Modified for Autism Spectrum Disorder (CYBOCS-ASD) Score
Description: The Children's Yale-Brown Obsessive Compulsive Scale modified for Autism Spectrum Disorder is a 5-item clinician-rated measure to evaluate severity of repetitive behavior in children with ASD. Each item is scored on a 5 point scale from 0 (None) to 4 (Extreme) for the severity of: Time Spent, Interference in everyday life, Distress, Resistance, and Degree of Control over the behavior. A total score ranges from 0 to 20. Lower scores are better.
Time Frame: Before (Baseline), After Part I (Week 12), After Part 2 (Week 24)
Measure: Mean (Standard Deviation); unit: Raw Score
Arm/Group | Wide-spectrum Nutritional Supplement | Placebo Control
Number analyzed (Participants) | 16 | 16
Raw Score
  Before | 12.5 (2.5) | 12.9 (2.4)
  After | 11.3 (2.3) | 11.9 (2.3)

8. Secondary Outcome: Change in the Aberrant Behavior Checklist (ABC) Scores
Description: The Aberrant Behavior Checklist is a 58-item caregiver questionnaire consisting of five subscales: hyperactivity, irritability, social withdrawal, stereotypic behavior and inappropriate speech in children with developmental disabilities. A higher score indicates more frequent aberrant behaviors. Our secondary measures are the subscale scores for Irritability (15 item), Social Withdrawal (16 item) and Hyperactivity (16 item). Each item rates behavior severity on a 4 point scale from 0 (Not at all a problem) to 3 (The problem is severe in degree). Total score ranges from 0 to 174. Lower scores are better.
Time Frame: Before (Baseline), After Part I (Week 12), After Part 2 (Week 24)
Measure: Mean (Standard Deviation); unit: Raw Score
Arm/Group | Wide-spectrum Nutritional Supplement | Placebo Control
Number analyzed (Participants) | 16 | 16
Raw Score
  Before | 77.136 (6.964) | 79.859 (6.964)
  After | 57.293 (6.964) | 73.87 (6.964)

9. Secondary Outcome: Change in the Parent-rated Anxiety Scale for ASD (PRAS-ASD) Score
Description: The Parent-rated Anxiety Scale for Autism Spectrum Disorder is a 25-item scale that measures anxiety in youth with ASD. Each item rates the severity of a behavior on a 4 point scale from 0 (None/not present) to 3 (Severe/Very frequent and a major problem). The total score ranges from 0 to 75. Lower scores are better.
Time Frame: Before (Baseline), After Part I (Week 12), After Part 2 (Week 24)
Measure: Mean (Standard Deviation); unit: Raw Score
Arm/Group | Wide-spectrum Nutritional Supplement | Placebo Control
Number analyzed (Participants) | 16 | 16
Raw Score
  Before | 30.25 (6.61) | 23.18 (6.61)
  After | 14.625 (6.61) | 26.1 (6.61)

10. Secondary Outcome: Change in the Caregiver Strain Questionnaire (CGSQ) Score
Description: The Caregiver Strain short-form questionnaire is a 7-item measure of self-reported strain experienced by caregivers of children with behavioral disorders. Each item rates the severity of interference in the quality of the caregiver's life on a 5 point scale from 0 (Not at All) to 4 (Very Much). The scale ranges from 0 to 28. Lower scores are better.
Time Frame: Before (Baseline), After Part I (Week 12), After Part 2 (Week 24)
Measure: Mean (Standard Deviation); unit: Raw Score
Arm/Group | Wide-spectrum Nutritional Supplement | Placebo Control
Number analyzed (Participants) | 16 | 16
Raw Score
  Before | 18.25 (2.695) | 17.625 (2.695)
  After | 11.5 (2.695) | 14.93 (2.695)

11. Secondary Outcome: Change in the Vineland III Caregiver Score
Description: The Vineland III Caregiver is a 381-item parent-reported measure of adaptive behavior in children with developmental and intellectual disabilities. The Vineland is comprised of three sub scores for the following domains: Communication, Daily Living Skills, and Socialization. The frequency of adaptive behaviors for each item is scored on a scale from 0 (Never) to 2 (Usually). The total adaptive score is reflected as a composite score of the sub domains (which is determined by age norms) in which a higher total score reflects higher functioning. The scale is standardized with a mean of 100 and standard deviation of 15.
Time Frame: Before (Baseline), After Part I (Week 12), After Part 2 (Week 24)
Measure: Mean (Standard Deviation); unit: Scaled Score
Arm/Group | Wide-spectrum Nutritional Supplement | Placebo Control
Number analyzed (Participants) | 16 | 16
Scaled Score
  Before | 62.645 (2.278) | 65.199 (2.278)
  After | 69.861 (2.278) | 62.175 (2.278)

12. Secondary Outcome: Evaluate Intervention Safety
Description: Columbia-Suicide Severity Rating Scale: a suicide risk assessment that identifies presence and severity of suicidal ideation, planning, and behavior, as well as non-suicidal self-harm behaviors. Presence of any of these behaviors during the course of study enrollment will be considered an adverse event.
Time Frame: Screening, Baseline, After Week 4, After Week 8, After Week 12, Atter Week 16, After Week 20, After Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Wide-spectrum Nutritional Supplement | Placebo Control
Number analyzed (Participants) | 16 | 16
Participants | 0 | 0

13. Secondary Outcome: Examine the Change in Cognitive Ability
Description: Differential Abilities Scale-II: cognitive abilities across core domains: verbal, nonverbal, spatial. Subtests: Verbal comprehension: 42-item domain, raw score 0-23. Naming vocabulary: 34-item domain, raw score 0-28. Word definitions: 35-item domain, raw score 0-25. Verbal similarities: 33-item domain, raw score 0-28. Picture similarities: 32-item domain, raw score 0-23. Picture similarities: 50-item domain, raw score 0-34. Matrices: 56-item domain, raw score 0-33. Pattern construction: 35-item domain, raw score 0-74. Copying: 20-item domain, raw score 0-36. Recall of designs: 22-item domain, raw score 0-43. All subdomains have a t-score range of 10-90. Verbal ability standard score ranges from 30-170. Nonverbal ability standard score ranges from 32-170. Spatial ability standard score ranges from 34-170. Total General Conceptual Ability standard score ranges from 30-170. Subtests and item sets given vary by participant age. Higher scores are better.
Time Frame: Before (Baseline), After Part I (Week 12), After Part 2 (Week 24)
Measure: Mean (Standard Deviation); unit: Scaled Score
Arm/Group | Wide-spectrum Nutritional Supplement | Placebo Control
Number analyzed (Participants) | 16 | 16
Scaled Score
  Before | 73.627 (5.177) | 65.488 (5.177)
  After | 76.764 (5.177) | 74.143 (5.177)

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Wide-spectrum Nutritional Supplement | Placebo Control
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 1/16 | 0/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Wide-spectrum Nutritional Supplement (N=16) | Placebo Control (N=16)
Mild transient constipation, diarrhea, and acid reflux (Gastrointestinal disorders) | 1 (1) | 0 (0) — Mild transient constipation, diarrhea, and acid reflux

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-11): https://cdn.clinicaltrials.gov/large-docs/17/NCT03835117/Prot_SAP_000.pdf